CLINICAL TRIAL: NCT06716281
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of IxCell hUC-MSC-O in Patients With Knee Osteoarthritis
Brief Title: Efficacy and Safety of IxCell hUC-MSC-O in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai IxCell Biotechnology Co., LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LC-MSCOA23001
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC group (Experimental): IxCell hUC-MSC-O;2.5×10^7 cells/1 mL, 1 mL/vial; 2ml
  Interventions: Biological: Human umbilical cord mesenchymal stem cells
- placebo group (Placebo Comparator): Sodium Chloride Injection；1 mL/vial；2ml
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — a single intra-articular injection of IxCell hUC-MSC-O at a dose of 5.0×10^7 cells with a volume of 2.0 mL
  Arms: MSC group
Biological: Placebo — Sodium Chloride Injection
  Arms: placebo group

SUMMARY:
To evaluate the efficacy of IxCell hUC-MSC-O in the treatment of patients with knee osteoarthritis.

To evaluate the safety of IxCell hUC-MSC-O in the treatment of patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs), as a kind of cells with multiple differentiation potential, have gradually shown their advantages in the treatment of osteoarthritis (OA) cartilage lesions. MSCs exist widely in connective tissues and interstitial organs of the whole body, such as bone marrow, umbilical cord, fat, etc., and can become specialized cells to perform functions under specific signal stimulation. MSCs can also secrete a variety of enzymes and nutritional factors such as growth factors, cytokines, chemokines, etc. to participate in the paracrine process, and play anti-apoptosis, anti-fibrosis, anti-oxidation, anti-inflammatory and pro-angiogenesis roles. In vitro studies and a number of clinical studies have confirmed that direct injection of MSCs into the joint cavity has a certain therapeutic effect on OA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with knee osteoarthritis according to the "Guidelines for the Diagnosis and Treatment of Osteoarthritis (2018 Edition)" by the Joint Surgery Group of the Orthopedics Branch of the Chinese Medical Association;
2. Patients with persistent pain for more than half a year, or those whose knee osteoarthritis recurs or worsens after discontinuing conventional clinical treatments such as hormones, opioids, non-steroidal anti-inflammatory drugs, viscosupplementary therapy, etc.;
3. The study side knee joint Kellgren-Lawrence grade is II～III, and the other side knee Kellgren-Lawrence is ≤II;
4. Patients with a total WOMAC score of ≥50 and ≤150 at the time of screening;
5. Patients with a VAS pain score of ≥50mm (total score of 100mm) in the study side knee joint at the time of screening;
6. Ages between 40 and 80, with no gender restrictions. BMI (Body Mass Index, weight [kg]/height^2 [m^2]) ≤30;
7. Able to understand and voluntarily sign the informed consent form, and willing to complete the trial procedures and follow-up examinations.

Exclusion Criteria:

1. Patients diagnosed with secondary knee osteoarthritis;
2. Patients with other diseases that cause knee joint dysfunction or affect the joint (such as acute joint injuries caused by trauma, rheumatoid arthritis, metabolic bone disease, psoriatic arthritis, gouty arthritis, symptomatic chondrocalcinosis, osteonecrosis, or active infections, lower limb arteriosclerosis obliterans, etc.);
3. Patients with obvious varus or valgus deformities (greater than 15 degrees) in the knee joint or with obvious flexion contractures;
4. Patients who have previously used stem cell therapy;
5. Patients who have received opioid, non-steroidal anti-inflammatory analgesics, or any other pain-relieving medication for knee osteoarthritis within 2 weeks or 7 half-lives (whichever is longer) before treatment;
6. Patients who have received physiotherapy or traditional Chinese medicine treatment for knee arthritis (either side) within 6 weeks before treatment;
7. Patients who have received local injection of glucocorticoids, anesthetics, or local application of glucocorticoids for the knee joint (either side) within 12 weeks before treatment, or who have received systemic glucocorticoid treatment within 12 weeks, or who require systemic glucocorticoid treatment during the study;
8. Patients who started taking glucosamine, chondroitin sulfate, or diacerein within 4 weeks before treatment (except those who have been taking glucosamine or chondroitin sulfate for a long time and have continued to take them for 4 weeks before treatment and are willing to maintain the dosage and frequency during the study);
9. Patients who have received any drug injection treatment in the knee joint cavity (either side) within 6 months before treatment;
10. Patients who have undergone major surgery, arthroplasty, or arthroscopy on the study side knee joint within 24 weeks before signing the informed consent form, or those who plan to undergo surgical treatment on the study side knee joint during the study;
11. Patients who have undergone surgical treatment on the lower limbs (hip or knee) within 12 weeks before signing the informed consent form;
12. Patients whose study side knee joint is not suitable for MRI examination, such as those with metal implants affected by magnetic fields;
13. Patients who plan to undergo any type of lower limb surgery within 48 weeks after signing the informed consent form;
14. Patients with skin diseases or skin infections around the intended injection site;
15. Patients with osteoarthritis on the opposite side of the study knee joint and who plan to undergo intra-articular drug therapy during the study;
16. Patients with hip joint disease on the same side as the study knee joint and who require medical intervention (such as severe hip osteoarthritis);
17. Patients with a history of allergic reactions to any components of the trial medication;
18. Patients with current malignant tumors or a history of malignant tumors within 5 years before signing the informed consent form;
19. Patients with a clear history of mental disorders, or a history of abuse of psychotropic drugs or drug use;
20. Patients with severe heart disease (NYHA Class III or above), or liver function abnormalities (serum ALT > 3×ULN or AST > 3×ULN), or kidney function abnormalities (serum Cr > 2×ULN or BUN > 2×ULN), or coagulation disorders (INR > 1.5), or severe hematological diseases (such as anemia of grade 3 or above, Hb < 8g/dL, or thrombocytopenia of grade 2 or above, Plt < 75×10^9/L);
21. Patients with HBeAg-positive chronic hepatitis B (defined by the 2015 Guidelines for the Prevention and Treatment of Chronic Hepatitis B), or hepatitis C virus infection, or positive for human immunodeficiency virus antibodies, or positive for Treponema pallidum antibodies;
22. Female patients who are pregnant or breastfeeding, or male and female patients who refuse to use contraceptive measures (abstinence, physical contraception, or hormonal contraceptives starting 3 months before enrollment) from the study period to 6 months after the last visit;
23. Patients who have participated in any other clinical trials within 3 months before signing the informed consent form;
24. Patients deemed unsuitable for participation in this trial by the investigator for other reasons.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
WOMAC total score | 48 week
  The change in WOMAC total score from baseline at 48 weeks post-dose.
cartilage damage | 48 week
  The change in cartilage damage area from baseline at 48 weeks post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhao, Principal Investigator — The Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- The Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China